CLINICAL TRIAL: NCT03320278
Title: Evaluation of the Effectiveness of Simplified Predictive Intubation Difficulty Score in Difficult Airway
Brief Title: The Evaluation of Simplified Predictive Intubation Difficulty Score.
Status: Completed | Type: Observational
Sponsor: Maltepe University (Other)
Collaborators: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Onur Selvi, assistant professor, Maltepe University
Other Study IDs: 2016/900/39
Record Dates: First submitted 2016-10-24; First posted 2017-10-25 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Head and Neck Disorder; Difficult Intubation; Facial Deformity
Keywords: endotracheal intubation; airway management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SPIDS,TMH: There will be two tests in this study for evaluation. Both of them will be measured in same group.

SUMMARY:
Difficult intubation is considered one of the most important obstacle increasing mortality in anesthesiology. Airway assessment tests are proceeded to overcome these difficulties in the pre-anesthetic evaluation. In this study, the Simplified Predictive Intubation Difficulty Score (SPIDS) and Thyromental Height Measurement (TMH) were chosen as primary methods to predict difficult intubation. The ear-nose-throat (ENT) and Plastic Surgery patients were planned to enroll this study to assess the effectiveness of these tests in predicting difficult intubation in Maltepe University Hospital and Sisli Hamidiye Etfal Governmental Hospital.

The SPIDS of volunteers will be calculated according to their previous knowledge of difficult intubation, airway pathologies, head and neck movements, mouth opening, modified Mallampati test and thyromental distance. TMH value will be measured with ASIMETO depth device. Finally, the SPIDS and TMH values will be statistically compared to predict difficult intubation which is determined with difficult intubation score (IDS).

DETAILED DESCRIPTION:
The investigators would like to evaluate consecutively patients, who applied to be operated in plastic surgery and ENT clinics due to head and neck pathologies which may cause difficult intubation, between May 2016 and December 2017 . The patients will be recruited to study consecutively therefore, there is going to be no randomization. The patients' height, age, weight, American Society of Anesthesiology (ASA) scores will be documented. Additionally, their Mallampati scores, thyromental distance, thyromental height, mouth opening values will be measured with ASIMETO DEPTH GAUGE digitally. Head and neck movement angle measurement will proceed in preoperative evaluation. In the operation room the intubation, determination of C-L and IDS are going to be operated by the anesthesiologist who is in charge of operating room and he or she will not be informed about airway assessments like SPIDS or TMH. The all difficult airway equipment will be readily prepared in advanced. Recorded data will be collected by the assistant researcher. The existing difficult intubation interventions will be determined by using IDS. The relationship between IDS, TMH and SPIDS values will be assessed in the means of predicting difficult airway.

Measurements:

Mallampati score: It has four grades and Mallampati 3 and 4 considered predictive factor for difficult intubation Thyromental distance (TMD): Short thyromental distance (TMD ≤ 6.5 cm) has been correlated with difficult direct laryngoscopic intubation in adult patients.

Thyromental height (TMH): This is a new technique for predicting difficult intubation and its accepted cut off is generally 5cm.

Height/Thyromental distance: Ratio of height in cm and thyromental distance in cm Intubation difficulty score (IDS): 0 is easy, 0-5 is slight difficulty and higher than 5 is moderate or serious difficulty in intubation.

The simplified descriptive intubation difficulty score (SPIDS): The maximum score can be 55 and the total score greater than 10,not SPIDS ≤ 10 is considered as difficult intubation. Calculation of SPIDS score following parameters is needed.

1. History of pathologies might be related to difficult intubation such as obstructive sleep apnea, facial malformations, cervical dislocation etc. no is 0, yes 10 is points
2. Mouth opening: ≥3.5 cm (0 points)- ≤3.5 cm (10 points)
3. Maximum head and neck measurement ≥80°(0 points), <80 (5 points)
4. Modified Mallampati test: class 1 (0 point ), class 2 (10 points), class 3 (15 points), class 4 (25 points)

ELIGIBILITY:
Inclusion Criteria:

* Being volunteer
* Older than 18 years old
* Being undergoing planned elective surgery patients
* Being ENT or plastic surgery patient

Exclusion Criteria:

* Emergency operations
* Patients younger than 18 years old
* Being non-volunteer for the study
* Patients will not be orally intubated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Volunteers in ENT and plastic surgery patients with possibly have maxillary,oral,head and neck pathologies
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
SPIDS | 6 months
  SPIDS - Simplified Predictive Intubation Difficulty Score - calculated using patient history, mouth opening, maximum angle of head and neck mobility and modified Mallampati test

SECONDARY OUTCOMES:
comparing sensitivity and specificity of TMH and SPIDS in predicting difficult airway | 6 months
  TMH with cut off value is 5cm is considered as a good predictor for difficult airway. SPIDS is greater than 10 is considered as difficult intubation. Comparing this two measurement techniques for predicting difficult intubations will be calculated with Receiver Operating characteristics (ROC) analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha Ozer, Prof., Study Chair — Maltepe University Medica Faculty
Locations (1):
- Maltepe University, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] L'Hermite J, Nouvellon E, Cuvillon P, Fabbro-Peray P, Langeron O, Ripart J. The Simplified Predictive Intubation Difficulty Score: a new weighted score for difficult airway assessment. Eur J Anaesthesiol. 2009 Dec;26(12):1003-9. doi: 10.1097/EJA.0b013e32832efc71. PMID 19593145
- [Result] Arne J, Descoins P, Fusciardi J, Ingrand P, Ferrier B, Boudigues D, Aries J. Preoperative assessment for difficult intubation in general and ENT surgery: predictive value of a clinical multivariate risk index. Br J Anaesth. 1998 Feb;80(2):140-6. doi: 10.1093/bja/80.2.140. PMID 9602574
- [Result] Etezadi F, Ahangari A, Shokri H, Najafi A, Khajavi MR, Daghigh M, Moharari RS. Thyromental height: a new clinical test for prediction of difficult laryngoscopy. Anesth Analg. 2013 Dec;117(6):1347-51. doi: 10.1213/ANE.0b013e3182a8c734. PMID 24257384
- See also: pubmed direct link — http://www.ncbi.nlm.nih.gov/pubmed